CLINICAL TRIAL: NCT00082303
Title: Music Imagery for Patients in Protected Environments
Brief Title: Music Imagery for Patients Receiving Chemotherapy for Leukemia or Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F32AT001144-01 (NIH)
Record Dates: First submitted 2004-05-05; First posted 2004-05-06 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Leukemia; Lymphoma, Non-Hodgkin
Keywords: Music Therapy; Anxiety; Depression
MeSH Terms: conditions — Leukemia; Lymphoma, Non-Hodgkin; Anxiety Disorders; Depression

INTERVENTIONS:
Behavioral: Music Imagery

SUMMARY:
The purpose of this study is to explore the effect of music imagery on patients receiving intensive chemotherapy for acute leukemia or high-grade non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
Standard treatment for acute leukemia and high-grade non-Hodgkin's lymphoma includes intensive chemotherapy that typically requires a 4-week hospital stay in protective isolation. Patients treated in isolation units may experience elevated levels of psychological distress. Both guided imagery and music therapy have been effective in improving the moods of cancer patients, but studies have not been conducted in acute leukemia and non-Hodgkin's lymphoma patients. This study will evaluate the effect of music imagery on these patients.

Participants in this study will be randomly assigned to receive either standard care plus music imagery or standard care alone. Participants assigned to the standard care plus music imagery group will receive a 45-minute weekly music imagery session with a music therapist. All participants will complete questionnaires and self-reports regarding their general anxiety, affect, and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Indiana University Hematologic Malignancy Program for the treatment of newly diagnosed or recurrent acute leukemia or high-grade non-Hodgkin's lymphoma
* Able to read and understand English

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2002-07

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Cancer Center/University Hospital, Indianapolis, Indiana, United States